CLINICAL TRIAL: NCT05255939
Title: Decrease Artery Occlusion by Distal Radial Arterial Cannulation in ACS Patients
Acronym: DONATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DONATION
Record Dates: First submitted 2022-01-17; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Acute Coronary Syndrome; Procedural Complication
Keywords: Distal Radial Access; Radial Artery Occlusion; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Acute Coronary Syndrome; Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dTRA group (Experimental): Investigators perform percutaneous coronary intervention by dTRA
  Interventions: Procedure: distal TRA group
- TRA group (Other): Investigators perform percutaneous coronary intervention by conventional TRA
  Interventions: Procedure: conventional TRA group

INTERVENTIONS:
Procedure: distal TRA group — dTRA for PCI procedure to ACS patients.
  Arms: dTRA group
Procedure: conventional TRA group — Conventional TRA for PCI procedure to ACS patients
  Arms: TRA group

SUMMARY:
The site of arterial access for coronary angiography and intervention has been the focus of research for decades as it is the source of major complications. Transradial access (TRA) reduces complications among patients undergoing percutaneous coronary procedures but is reported with the complication of radial artery occlusion (RAO) that limits the radial artery for future needs.

Distal radial access (dTRA) has recently gained global popularity as an alternative access route for vascular procedures. Among the benefits of dTRA are the low risk of entry site bleeding complications, the low rate of radial artery occlusion, and improved patient and operator comfort.

This study aims to reveal the feasibility and safety of dTRA and routine TRA procedures in acute coronary syndrome patients. The primary endpoints are forearm radical occlusion rate and major adverse cardiovascular events (MACEs) in the two groups, respectively. Investigators will also focus on puncture success in diagnostic and interventional cases, rate of One attempt success, access time, procedure time, crossover rate, contrast dose of patients, fluoroscopy time and dose, and healthcare cost of each group.

ELIGIBILITY:
Inclusion Criteria:

* presence of a pulse in the snuffbox

Exclusion Criteria:

* Absence of pulse
* Ultrasound indication of arterial occlusion or severe calcification
* Severe forearm artery malformation
* Patients with severe liver and renal failure, or abnormal coagulation function
* Established cardiogenic shock
* History of previous coronary artery bypass grafting and radial artery use.
* Raynaud's disease in the medical history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Forearm radical occlusion | during procedure
  Doppler ultrasound to determine whether patients suffer forearm radial occlusion
MACEs | during procedure
  Major Adverse Cardiovascular Events, including cardiovascular death, myocardial infarction and heart failure.

SECONDARY OUTCOMES:
Rate of One attempt success | during procedure
  Rate of One attempt success of 2 kinds of procedure
Access time | during procedure
  Access time of 2 kinds of procedure
Procedure time | during procedure
  Procedure time of 2 kinds of procedure
Crossover rate | during procedure
  Crossover rate of 2 kinds of procedure
Contrast dose | during procedure
  Contrast dose of 2 kinds of procedure
Fluoroscopy dose | during procedure
  Fluoroscopy dose of 2 kinds of procedure
hand hematoma | during procedure
  hand hematoma rate of 2 kinds of procedure
The total cost in hospitalization | up to 2 years
  Healthcare cost .

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No